CLINICAL TRIAL: NCT05393388
Title: Tau Pet Imaging in the Aging Brain Cohort Dedicated to Diversity Study
Acronym: ABCD2-TAU
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 844403
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Decline; Alzheimer Disease
Keywords: Healthy Subjects
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PET/CT: PET.CT using the radiotracer [18F]AV-1451
  Interventions: Drug: [18F]AV-1451

INTERVENTIONS:
Drug: [18F]AV-1451 — [18F]AV-1451 has been developed as a positron emitting radiopharmaceutical for in vivo imaging of tau protein aggregates.
  Other Names: [F-18]T807

SUMMARY:
We will conduct a Tau PET scan in cognitively normal older adults, enrolled in the Aging Brain Cohort Dedicated to Diversity Study (ABCD2-Tau) study at the University of Pennsylvania's Penn Memory Center/Alzheimer's Disease Core Center (PMC/ADC).Study duration will generally be a one-day study visit for PET imaging, but all subjects will be followed annually as part of their participation in the ABCD2 study. Findings from this study will likely provide insight into the mechanisms and distinctions of age-related cognitive decline and that of preclinical Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females African Americans ≥ 65 years of age.
2. Part of the ABCD2 longitudinal cohort, protocol 844047, of the PMC/ADCC with consensus conference designation of normal cognition.
3. ABCD2 longitudinal visit must be completed or scheduled to be completed within 1 year prior to the [18F]AV-1451 TAU PET scan.
4. A brain MRI must be performed within 1 year prior to their study [18F]AV-1451 TAU PET scan date and be deemed of adequate quality that the scan may be used for study analysis, including 3T high-resolution imaging of medial temporal lobe structures.
5. An amyloid PET scan completed or scheduled within 1year of their study [18F]AV-1451
6. Women must be post-menopausal or surgically sterile.

Exclusion Criteria:

1. Have any medical or psychiatric conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study, including major depression and prior head trauma.
2. Have evidence of structural abnormalities such as major stroke or mass on MRI that is likely to interfere with analysis of the PET scan.
3. Inability to tolerate or contraindication to imaging procedures in the opinion of an investigator or treating physician.
4. Have a history of significant ongoing alcohol or substance abuse or dependence based on self-report.
5. Women of child bearing potential

   * The inclusion / exclusion criteria will be ascertained through self-report in conjunction with any medical history available through the participant's medical or research records (EPIC or the ADC database)*

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Study population includes cognitively normal, older adult (>65 years old) black or African American participants
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Uptake of [18F]AV-1451 in the medial temporal lobe | 4 years
  A quantitative measurement of [18F]AV-1451(standardized value uptake ratio - SUVR) within the medial temporal lobe (MTL).from PET/CT
Volume of medial temporal lobe subregion | 4 years
  A quantitative measurement of volume (milimeters - mm) of medial temporal lobe (MTL) subregion from a high resolution MRI.
Thickness of medial temporal lobe subregion | 4 years
  A quantitative measurement of thickness (milimeters - mm) of medial temporal lobe (MTL) subregion from a high resolution MRI.

CONTACTS AND LOCATIONS:
Overall Officials: David A Wolk, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania - Penn Memory Center, Philadelphia, Pennsylvania, United States